CLINICAL TRIAL: NCT06758154
Title: Efficacy and Olfactory Network of Electro-acupuncture for Subjective Cognitive Decline: A Multicenter Randomized Controlled Trial and fMRI Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-050-01
Record Dates: First submitted 2024-12-25; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-01

CONDITIONS: Subjective Cognitive Decline (SCD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Device: "TXJN" electro-acupuncture
- Control group (Sham Comparator)
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: "TXJN" electro-acupuncture — Firstly, EA treatment will be administered at the Neiguan (PC6, bilateral), Shenting(GV23), Yingxiang(LI20, bilateral), Yintang(GV29) acupoints. Disposable stainless-steel needles (0.25 mm × 25 mm; Huatuo brand, Suzhou Medical Supplies Factory Co., LTD., Suzhou City, China) will be used. After skin disinfection, the acupuncturists will twist and thrust the needle handles to achieve the sensations of achiness, heaviness, and numbness (known as de qi) at all above-mentioned acupoints. Following needle manipulations, EA instruments (SDZ-V, Hwato brand, Suzhou Medical Supplies Factory Co., Ltd., Suzhou City, China) will be used to attach the needle handles at PC6, GV23, LI20, GV29, with a dilatational wave of 5 Hz and a current intensity of 2 ~ 4 mA depending on the patient's tolerance. The needles will be removed after 30 min. Participants will receive 24 sessions over 8 weeks at a frequency of 3 times per week.
  Arms: Experimental group
Device: sham acupuncture — Firstly, EA treatment will be administered at the non-acupoints near above-mentioned real acupoints. Disposable stainless-steel needles (0.25 mm × 25 mm; Huatuo brand, Suzhou Medical Supplies Factory Co., LTD., Suzhou City, China) will be used. After skin disinfection, the acupuncturists will take the needle into the acupoints without the sensations of de qi. Following needle manipulations, EA instruments (SDZ-V, Hwato brand, Suzhou Medical Supplies Factory Co., Ltd., Suzhou City, China) will be used to attach the needle handles at non-acupoints without the current. The needles will be removed after 30 min. Participants will receive 24 sessions over 8 weeks at a frequency of 3 times per week.
  Arms: Control group

SUMMARY:
Subjective cognitive decline (SCD) is the early diagnosis and treatment window period of Alzheimer's disease (AD), and the identification of SCD individuals who will progress to AD (pSCD) is a research hotspot. Based on olfactory fMRI,previous studies have found that SCD individuals showed damaged entorhinal neural circuits. After follow-up, the incidence of pSCD increased by three times. But,the spatiotemporal characteristics of the entorhinal neural circuits and whether it has the value of individualized prediction and intervention target need to be further studied. Thus, based on multi-center ambispective cohort study at home and abroad, we will (1) build a new paradigm of synchronous fMRI-EEG olfactory task state Oddball experiment, jointly representational similarity analysis, extract spatiotemporal characteristics of neural circuits damage, and discover and verify that the entorhinal neural circuits are vulnerable brain regions; (2) establish the middle fusion model of vulnerable brain region combined with the methods of olfactory task-fMRI activation image generation, functional connectome gradient,etc.; Then, establish late fusion multi-omics multi-task model combined with the new methods of molecularomics such as ultra-deep total proteomics and metabonomics proposed by the research group to accurately identify pSCD; (3) carry out the precise intervention of image-guided "olfactory three-needle" acupuncture with the entorhinal neural circuits as the target. Through clinical RCT research and mouse model, the remodeling mechanism of vulnerable brain regions will be clarified.This project will provide the basis for early diagnosis and treatment of the AD risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for SCD diseases;
2. 55-79 years old;
3. ≥8 years of schooling;
4. Right-handed;
5. Sign the informed consent.

Exclusion Criteria:

1. Have received other antidepressant therapy or involved in other clinical trials in the previous 2weeks.
2. Infarct located in the left DLPFC.
3. Positive psychiatric history and major trauma exposure history, such as depression, epilepsy, etc., in the past.
4. Other serious concomitant diseases (aphasia, severe edema, venous thrombosis, arteriosclerosis occlusion, diabetic vascular disease, peripheral neuropathy, spinal lesions, brain trauma, intracranial infection, brain tumors, etc.) or secondary diseases (heart, liver, renal failure, etc.).
5. Infection around acupoints and/or intolerance to acupuncture manipulation.
6. MRI or rTMS contraindications (claustrophobia, metal implants, cochlear implants, impulsator, etc.).

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Z score | Before and 8 weeks after treatment
  The neuropsychological scale of 8 objective cognitive assessments used in the study (including AVLT (S and L), AFT, BNT, TMT (A and B), SCWT-C, DSST, DST, CDT) was converted into Z scores for description. Specific operations: Standardize the score of a single cognitive domain scale, create the corresponding Z-score data set, calculate the average value of each data in the group to generate a single Z-score, and sum the Z-score of each single cognitive domain to generate the overall Z-score. Patients were evaluated before treatment and 8 weeks later.
Multimodal magnetic resonance imaging of olfactory related neural circuits | Before and 8 weeks after treatment
  Structural MRI(3DTIWI/3DT2WI/3Dflair), functional MRI(BOLD\NODDI\ASL\ QSM)

SECONDARY OUTCOMES:
mini-mental state examination, MMSE | Before and 8 weeks after treatment
Montreal Cognitive Assessment,MoCA | Before and 8 weeks after treatment
Subjective cognitive self-scoring | Before and 8 weeks after treatment
Hamilton Depression Scale，HAMD | Before and 8 weeks after treatment
the Geriatric Depression Scale,GDS | Before and 8 weeks after treatment
Hamilton Anxiety Scale,HAMA | Before and 8 weeks after treatment
auditory verbal learning test,AVLT | Before and 8 weeks after treatment
Rey complex figure test,CFT | Before and 8 weeks after treatment
Boston naming test,BNT | Before and 8 weeks after treatment
Animal fluency test,AFT | Before and 8 weeks after treatment
rail making test-A,TMT-A | Before and 8 weeks after treatment
rail making test-B,TMT-B | Before and 8 weeks after treatment
complex figure test, CFT | Before and 8 weeks after treatment
clock drawing test,CDT | Before and 8 weeks after treatment
Symbol Digit Modalities Test,SDMT | Before and 8 weeks after treatment
odor threshold test,OTT | Before and 8 weeks after treatment
The olfactory behavioral test | Before and 8 weeks after treatment
Spatial navigation behavior test | Before and 8 weeks after treatment
Pittsburgh sleep quality index,PSQI | Before and 8 weeks after treatment
TCM physique classification scale | Before and 8 weeks after treatment
TCM syndrome type scale of mild cognitive impairment | Before and 8 weeks after treatment

OTHER OUTCOMES:
Acceptance survey | After 8 weeks of treatment
Adverse event | During treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR